CLINICAL TRIAL: NCT01222962
Title: Study of the Effect of Food on the Pharmacokinetics of DHA and PQP After Single Oral Administration of Eurartesim™ in Healthy Male Adult Volunteers
Brief Title: Food Interaction Study on the Pharmacokinetics of Eurartesim™ (DHA and PQP)in Healthy Male Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Giovanni Valentini, MD, Medical Department, R&D Division, Sigma-Tau ifr SpA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST3073/ST3074-DM09-008
Record Dates: First submitted 2010-10-11; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fed treatment (Experimental): 18 healthy volunteers administered with a single dose of Eurartesim
  Interventions: Drug: Eurartesim
- Fasted Treatment (Experimental): 18 healthy volunteers treated with a single dose of Eurartesim
  Interventions: Drug: Eurartesim

INTERVENTIONS:
Drug: Eurartesim — Tablet containing 40 mg of Dihydroartemisinin (DHA) and 320 mg of Piperaquine phosphate (PQP). 4 Tablets a Day for body weight above 75 kg.

SUMMARY:
The study was designed to assess the effect of food on the extent and rate of absorption of Dihydroartemisinin (DHA) and Piperaquine Phosphate (PQP) administered as a fixed dose combination (Eurartesim™).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian healthy males aged between 18 and 50 years(inclusive).
* Body Mass Index (BMI) between 19.0 kg/m2 and 27.0 kg/m2 inclusive, with a minimum body weight of 75 kg.
* Agreed to use two approved methods of contraception from Screening and until 90 days after administration of the study drug
* Had given written informed consent to participate in this study in accordance with local regulations.

Exclusion Criteria:

* Had received or was anticipated to receive a prescription medication within 14 days prior to the start of dosing or an over-the-counter medicine 48 hours prior to the start of dosing.
* Abnormal laboratory test results deemed clinically significant by the Medical Officer.
* Positive urine drug test (e.g. opiates and cannabinoids) or alcohol breath test.
* History of significant drug allergies or significant allergic reaction.
* Receipt of blood or blood products, or loss or donation of 450 mL or more of blood within 90 days before the first dose administration.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
tmax, Cmax, AUC0-last, AUC0-24 [PQ], and AUC0-inf, λz, t1/2, Cl/F, Vz/F [DHA]. | from the day of study drug administration, till Day 7 follow-up
  Blood samples for determination of plasma DHA were collected at the following times: At pre-dose Day 0 and then at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose.
  Blood samples for determination of plasma PQ were collected at the following times: At pre-dose Day 0 and then at 1, 2, 3, 4, 5, 6, 8, and 12 hours post-dose; on Day 1, 2, 3, 4, 5 and 7.

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events | Day 0 and till Day 30 follow-up
  Number of TEAEs and number of Subjects experiencing Adverse Events during all the study period
Hematology and blood chemistry changes respect to baseline values | Day 0, day 2, day 30
  Abnormalities in hematology (Haemoglobin, Hematocrit,RBC count, White cell count and differential count, Platelets) and clinical chemistry (Protein, Sodium, Potassium, Chloride ,Total Bilirubin, Conjugated Bilirubin, Alanine Aminotransferase, Aspartate Aminotransferase, Total Cholesterol, Glucose, Bicarbonate, Urea, Urate, Lactate Dehydrogenase, Albumin, Globulins, Triglycerides, Creatinine, Alkaline Phosphatase, Gamma glutamyltransferase, Total Calcium, Phosphate, C-reactive protein) will be recorded the day of the last study drug intake and after 30 days from the start of the drug treatment
QTc interval prolongation | Day 0, day 2, day 30
  ECG recordings will be obtained at baseline, after the last drug intake and 30 days follow-up to investigate changes in ECG parameters, and specifically QTc interval changes respect to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, a division of IDT Australia Limited, Adelaide, Australia